CLINICAL TRIAL: NCT00538629
Title: NON INTERVENTIONAL STUDY (NIS) IN PATIENTS WITH BIPOLAR DISCORDER (MANIC OR MIXED EPISODES) AND SCHIZOPHRENIA UNDERGOING TREATEMENT WITH ZELDOX
Brief Title: Non Interventional Study In Bipolar Disorder And Schizophrenia With Zeldox
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281171
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- schizophrenic: patients with schizophrenia
  Interventions: Other: no intervention
- bipolar disorder: patients with bipolar disorder
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: schizophrenic
Other: no intervention — no intervention
  Groups: bipolar disorder

SUMMARY:
Investigation of the impact of Zeldox on metabolic parametres in patients with bipolar disorder or with schizophrenia and impact of the treatment for the quality of life

DETAILED DESCRIPTION:
observational survey consecutive patient sampling

ELIGIBILITY:
Inclusion Criteria:

Manic and mixed episodes of up to moderate severity in patients with type I and II bipolar disorder and schizophrenia; either first diagnosed or repeated episodes.

Exclusion Criteria:

Patients with a history of hypersenzitivity to Ziprasidone. Previous insufficiency of the Ziprasidone´s treatment. The break of the previous therapeutic condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: psychiatric outpatients
Sampling Method: Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2007-10-16 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281171&StudyName=Non%20Interventional%20Study%20In%20Bipolar%20Disorder%20And%20Schizophrenia%20With%20Zeldox

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects enrolled had to have taken at least 1 dose of 40, 60, or 80 milligrams of ziprasidone. The study included subjects with diagnosed Type I or II bipolar disorder with manic and mixed episodes (n=223) and subjects with schizophrenia of up to moderate severity, either first diagnosed or repeated episodes (n=248).
Groups:
- Ziprasidone: Subjects had to have taken at least 1 dose of ziprasidone 40, 60, or 80 milligrams
Period: Overall Study
Arm/Group | Ziprasidone
Started | 471
Completed | 449
Not Completed | 22
Not completed — At subject's request | 1
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 6
Not completed — Subject's untimely distrust of medicine | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 471
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 2
  18-44 years | 294
  45-64 years | 152
  >=65 years | 23
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 198
  Female | 271
  Unspecified | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression of Severity (CGI-S) Scores (Bipolar Population)
Description: CGI-S assesses the severity of the condition at baseline using a scale that ranges from (1)Normal, not ill at all to (7) Among the most severely ill patients.
Time Frame: Baseline
Population: The bipolar full analysis set included all subjects with a diagnosis of bipolar mania who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  (1) Normal, not ill | 3
  (2) Borderline mentally ill | 5
  (3) Mildly ill | 19
  (4) Moderately ill | 57
  (5) Absolutely clearly ill | 101
  (6) Severely ill | 24
  (7) Among the most extremely ill subjects | 0
  Missing | 13

2. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Mental Health?
Description: MANSA is a 16-item self-assessment of satisfaction with quality of life. Items are rated on a 7-point scale, with higher score indicating greater satisfaction.
Time Frame: Baseline and final visit (week 12)
Population: The schizophrenia full analysis set included all subjects with a diagnosis of schizophrenia who had received at least 1 dose of study medication. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 176
Participants
  Baseline: Could not be worse | 13
  Baseline: Displeased | 45
  Baseline: Mostly dissatisfied | 36
  Baseline: Mixed | 44
  Baseline: Mostly satisfied | 19
  Baseline: Pleased | 17
  Baseline: Could not be better | 2
  Baseline: Missing | 68
  Final: Could not be worse: number analyzed (Participants) | 174
  Final: Could not be worse | 2
  Final: Displeased: number analyzed (Participants) | 174
  Final: Displeased | 20
  Final: Mostly dissatisfied: number analyzed (Participants) | 174
  Final: Mostly dissatisfied | 23
  Final: Mixed: number analyzed (Participants) | 174
  Final: Mixed | 54
  Final: Mostly satisfied: number analyzed (Participants) | 174
  Final: Mostly satisfied | 48
  Final: Pleased: number analyzed (Participants) | 174
  Final: Pleased | 26
  Final: Could not be better: number analyzed (Participants) | 174
  Final: Could not be better | 1
  Final: Missing: number analyzed (Participants) | 174
  Final: Missing | 70

3. Primary Outcome: Young Mania Rating Scale (YMRS) Scores (Bipolar Population): Change From Baseline
Description: The YMRS is an 11-item questionnaire that rates the severity of bipolar disorder, with higher score indicating greater severity of disease. Change: score at final visit minus score at baseline.
Time Frame: Baseline to final visit (12 weeks)
Population: The bipolar full analysis set included all subjects with a diagnosis of bipolar mania who had received at least 1 dose of study medication. If the final visit measurement was missing, the follow-up measurement could be carried forward. If any individual item was missing, the total score was set to missing. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 208
Score on scale
  Baseline | 26.6 (12.6)
  Final visit: number analyzed (Participants) | 207
  Final visit | 10.8 (8.3)
  Change from baseline | -15.6 (9.4)

4. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) Scores (Bipolar Population): Change From Baseline
Description: MADRS measures treatment effect on depression severity. MADRS assesses apparent and reported sadness, inner tension, sleep, appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Higher score indicates greater severity of disease. Change: score at final visit minus score at baseline.
Time Frame: Baseline to final visit (12 weeks)
Population: The bipolar full analysis set included all subjects with a diagnosis of bipolar mania who had received at least 1 dose of study medication. If any individual item was missing, the total score was set to missing. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 214
Score on scale
  Baseline | 26.2 (20.3)
  Final visit | 11.6 (9.1)
  Change from baseline: number analyzed (Participants) | 213
  Change from baseline | -14.6 (16.1)

5. Primary Outcome: Clinical Global Impressions Change (CGI-C) Scores (Bipolar Population)
Description: CGI-C assesses change in severity of the conditionusing a scale that ranges from (1) very much improved to (7) very much worse. Higher score indicates increasing severity of disease.
Time Frame: Final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  (1) Very much improved | 40
  (2) Much improved | 117
  (3) Minimally improved | 52
  (4) No change | 5
  (5) Minimally worse | 1
  (6) Much worse | 3
  (7) Very much worse | 0
  Missing | 4

6. Primary Outcome: Clinical Global Impressions Change (CGI-C) Scores (Schizoprenia Population)
Description: as for outcome 5
Time Frame: Final visit (week 12)
Population: The schizophrenia full analysis set included all subjects who had been diagnosed with schizophrenia and had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  (1) Very much improved | 22
  (2) Much improved | 125
  (3) Minimally improved | 76
  (4) No change | 14
  (5) Minimally worse | 1
  (6) Much worse | 3
  (7) Very much worse | 0
  Missing | 3

7. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Scores (Schizophrenia Population): Change From Baseline
Description: BPRS is an 18-item scale with 11 general symptom items, 5 positive-symptom items, and 2 negative symptom items. The physician completes the BPRS, and each item is scored on a 7-point scale, with higher score indicating greater severity of symptom. Change: score at final visit minus score at baseline.
Time Frame: Baseline to final visit (week 12)
Population: The schizophrenia full analysis set included all subjects with a diagnosis of schizophrenia who had received at least 1 dose of study medication. If any individual item was missing, the total score was set to missing. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 205
Score on scale
  Baseline | 49.3 (17.9)
  Final visit: number analyzed (Participants) | 165
  Final visit | 35.2 (11.3)
  Change from baseline: number analyzed (Participants) | 160
  Change from baseline | -20.0 (13.4)

8. Primary Outcome: Extrapyramidal Symptom (EPS) Scores (Schizophrenia Population: Baseline and Final Visit
Description: EPS assesses 4 items: akathisia, dystonia, dyskinesia, and parkinsonism. Each item is scored on a 5-point severity scale ranging from 1 to 5, with higher score indicating greater severity of symptom. Change: score at final visit minus score at baseline.
Time Frame: Baseline and final visit (week 12)
Population: The schizophrenia full analysis set included all subjects with a diagnosis of schizophrenia who had received at least 1 dose of study medication. If any individual item was missing, the total score was set to missing.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Score on scale
  Baseline: number analyzed (Participants) | 206
  Baseline | 7.0 (4.7)
  Final visit: number analyzed (Participants) | 213
  Final visit | 4.4 (2.9)

9. Primary Outcome: Global Efficacy Evaluation Scores (Bipolar Population)
Description: The Global Efficacy Evaluation assesses the final efficacy of ziprasidone on bipolar symptoms using a 5-point scale that ranges from very good to worsening of the original disease.
Time Frame: Final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Very good | 154
  Good | 24
  Average | 36
  Poor | 4
  Worsening of the original disease | 1
  Missing | 3

10. Primary Outcome: Global Efficacy Evaluation Scores (Schizophrenia Population)
Description: The Global Efficacy Evaluation assesses the final efficacy of ziprasidone on schizophrenia symptoms using a 5-point scale that ranges from very good to worsening of the original disease.
Time Frame: Final visit (week 12)
Population: The schizophrenia full analysis set included all subjects with a diagnosis of schizophrenia who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Very good | 166
  Good | 28
  Average | 35
  Poor | 7
  Worsening of the original disease | 3
  Missing | 5

11. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Life as a Whole Today?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 8
  Baseline: Displeased | 27
  Baseline: Mostly dissatisfied | 26
  Baseline: Mixed | 25
  Baseline: Mostly satisfied | 29
  Baseline: Pleased | 29
  Baseline: Could not be better | 11
  Baseline: Missing | 67
  Final: Could not be worse | 2
  Final: Displeased | 10
  Final: Mostly dissatisfied | 18
  Final: Mixed | 28
  Final: Mostly satisfied | 56
  Final: Pleased | 36
  Final: Could not be better | 3
  Final: Missing | 69

12. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Job?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 5
  Baseline: Displeased | 28
  Baseline: Mostly dissatisfied | 28
  Baseline: Mixed | 22
  Baseline: Mostly satisfied | 33
  Baseline: Pleased | 33
  Baseline: Could not be better | 6
  Baseline: Missing | 67
  Final: Could not be worse | 0
  Final: Displeased | 13
  Final: Mostly dissatisfied | 21
  Final: Mixed | 32
  Final: Mostly satisfied | 47
  Final: Pleased | 38
  Final: Could not be better | 1
  Final: Missing | 70

13. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Financial Situation?
Description: MANSA is a 16-item self-assessment of satisfaction with quality of life. Items are rated on a 7-point scale, with higher number indicating higher satisfaction.
Time Frame: Baseline and final visit (week 12)
Population: The bipolar full analysis set included all subjects who had been diagnosed with bipolar mania and had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 9
  Baseline: Displeased | 48
  Baseline: Mostly dissatisfied | 37
  Baseline: Mixed | 17
  Baseline: Mostly satisfied | 21
  Baseline: Pleased | 14
  Baseline: Could not be better | 5
  Baseline: Missing | 71
  Final: Could not be worse | 1
  Final: Displeased | 33
  Final: Mostly dissatisfied | 41
  Final: Mixed | 24
  Final: Mostly satisfied | 24
  Final: Pleased | 24
  Final: Could not be better | 1
  Final: Missing | 74

14. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: Do You Have Anyone You Would Call a Close Friend?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Yes | 112
  Baseline: No | 41
  Baseline: Missing | 69
  Final: Yes | 113
  Final: No | 37
  Final: Missing | 72

15. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: In the Last Week Have You Seen a Friend?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Yes | 88
  Baseline: No | 66
  Baseline: Missing | 68
  Final: Yes | 95
  Final: No | 54
  Final: Missing | 73

16. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With the Number and Quality of Your Friendships?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 2
  Baseline: Displeased | 32
  Baseline: Mostly dissatisfied | 22
  Baseline: Mixed | 27
  Baseline: Mostly satisfied | 34
  Baseline: Pleased | 29
  Baseline: Could not be better | 9
  Baseline: Missing | 67
  Final: Could not be worse | 1
  Final: Displeased | 18
  Final: Mostly dissatisfied | 24
  Final: Mixed | 26
  Final: Mostly satisfied | 43
  Final: Pleased | 40
  Final: Could not be better | 0
  Final: Missing | 70

17. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Accomodation?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 3
  Baseline: Displeased | 19
  Baseline: Mostly dissatisfied | 17
  Baseline: Mixed | 17
  Baseline: Mostly satisfied | 39
  Baseline: Pleased | 50
  Baseline: Could not be better | 7
  Baseline: Missing | 70
  Final: Could not be worse | 0
  Final: Displeased | 16
  Final: Mostly dissatisfied | 11
  Final: Mixed | 18
  Final: Mostly satisfied | 48
  Final: Pleased | 53
  Final: Could not be better | 0
  Final: Missing | 76

18. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Leisure Activities?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 4
  Baseline: Displeased | 28
  Baseline: Mostly dissatisfied | 29
  Baseline: Mixed | 19
  Baseline: Mostly satisfied | 31
  Baseline: Pleased | 31
  Baseline: Could not be better | 13
  Baseline: Missing | 67
  Final: Could not be worse | 0
  Final: Displeased | 13
  Final: Mostly dissatisfied | 24
  Final: Mixed | 26
  Final: Mostly satisfied | 49
  Final: Pleased | 40
  Final: Could not be better | 0
  Final: Missing | 70

19. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: In the Past Year Have You Been Accused of a Crime?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Yes | 7
  Baseline: No | 146
  Baseline: Missing | 69
  Final: Yes | 6
  Final: No | 143
  Final: Missing | 73

20. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: In the Past Year, Have You Been a Victim of Physical Violence?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Yes | 10
  Baseline: No | 144
  Baseline: Missing | 68
  Final: Yes | 9
  Final: No | 141
  Final: Missing | 72

21. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Personal Safety?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 1
  Baseline: Displeased | 14
  Baseline: Mostly dissatisfied | 12
  Baseline: Mixed | 35
  Baseline: Mostly satisfied | 37
  Baseline: Pleased | 50
  Baseline: Could not be better | 6
  Baseline: Missing | 67
  Final: Could not be worse | 2
  Final: Displeased | 6
  Final: Mostly dissatisfied | 6
  Final: Mixed | 21
  Final: Mostly satisfied | 54
  Final: Pleased | 58
  Final: Could not be better | 6
  Final: Missing | 69

22. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With the People You Live With?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 0
  Baseline: Displeased | 17
  Baseline: Mostly dissatisfied | 17
  Baseline: Mixed | 28
  Baseline: Mostly satisfied | 38
  Baseline: Pleased | 47
  Baseline: Could not be better | 7
  Baseline: Missing | 68
  Final: Could not be worse | 0
  Final: Displeased | 8
  Final: Mostly dissatisfied | 15
  Final: Mixed | 19
  Final: Mostly satisfied | 48
  Final: Pleased | 59
  Final: Could not be better | 3
  Final: Missing | 70

23. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Sex Life?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 11
  Baseline: Displeased | 41
  Baseline: Mostly dissatisfied | 17
  Baseline: Mixed | 32
  Baseline: Mostly satisfied | 15
  Baseline: Pleased | 29
  Baseline: Could not be better | 10
  Baseline: Missing | 67
  Final: Could not be worse | 6
  Final: Displeased | 28
  Final: Mostly dissatisfied | 22
  Final: Mixed | 27
  Final: Mostly satisfied | 34
  Final: Pleased | 36
  Final: Could not be better | 0
  Final: Missing | 69

24. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Relationship With Your Family?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 2
  Baseline: Displeased | 17
  Baseline: Mostly dissatisfied | 17
  Baseline: Mixed | 43
  Baseline: Mostly satisfied | 31
  Baseline: Pleased | 38
  Baseline: Could not be better | 7
  Baseline: Missing | 67
  Final: Could not be worse | 0
  Final: Displeased | 6
  Final: Mostly dissatisfied | 12
  Final: Mixed | 29
  Final: Mostly satisfied | 50
  Final: Pleased | 55
  Final: Could not be better | 1
  Final: Missing | 69

25. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Health?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 7
  Baseline: Displeased | 13
  Baseline: Mostly dissatisfied | 15
  Baseline: Mixed | 22
  Baseline: Mostly satisfied | 39
  Baseline: Pleased | 50
  Baseline: Could not be better | 9
  Baseline: Missing | 67
  Final: Could not be worse | 1
  Final: Displeased | 11
  Final: Mostly dissatisfied | 9
  Final: Mixed | 22
  Final: Mostly satisfied | 49
  Final: Pleased | 60
  Final: Could not be better | 1
  Final: Missing | 69

26. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Bipolar Population) in Answer to: How Satisfied Are You With Your Mental Health?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 222
Participants
  Baseline: Could not be worse | 6
  Baseline: Displeased | 29
  Baseline: Mostly dissatisfied | 19
  Baseline: Mixed | 32
  Baseline: Mostly satisfied | 18
  Baseline: Pleased | 35
  Baseline: Could not be better | 15
  Baseline: Missing | 68
  Final: Could not be worse | 0
  Final: Displeased | 9
  Final: Mostly dissatisfied | 17
  Final: Mixed | 34
  Final: Mostly satisfied | 45
  Final: Pleased | 45
  Final: Could not be better | 3
  Final: Missing | 69

27. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Life as a Whole Today?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 13
  Baseline: Displeased | 48
  Baseline: Mostly dissatisfied | 37
  Baseline: Mixed | 43
  Baseline: Mostly satisfied | 30
  Baseline: Pleased | 6
  Baseline: Could not be better | 0
  Baseline: Missing | 67
  Final: Could not be worse | 0
  Final: Displeased | 21
  Final: Mostly dissatisfied | 23
  Final: Mixed | 48
  Final: Mostly satisfied | 69
  Final: Pleased | 14
  Final: Could not be better | 0
  Final: Missing | 69

28. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Job?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 5
  Baseline: Displeased | 36
  Baseline: Mostly dissatisfied | 40
  Baseline: Mixed | 39
  Baseline: Mostly satisfied | 33
  Baseline: Pleased | 22
  Baseline: Could not be better | 0
  Baseline: Missing | 69
  Final: Could not be worse | 1
  Final: Displeased | 23
  Final: Mostly dissatisfied | 36
  Final: Mixed | 33
  Final: Mostly satisfied | 53
  Final: Pleased | 27
  Final: Could not be better | 0
  Final: Missing | 71

29. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores(Schizophrenia Population) in Answer to: How Satisfied Are You With Your Financial Situation?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 8
  Baseline: Displeased | 70
  Baseline: Mostly dissatisfied | 39
  Baseline: Mixed | 23
  Baseline: Mostly satisfied | 18
  Baseline: Pleased | 13
  Baseline: Could not be better | 1
  Baseline: Missing | 72
  Final: Could not be worse | 1
  Final: Displeased | 40
  Final: Mostly dissatisfied | 54
  Final: Mixed | 35
  Final: Mostly satisfied | 20
  Final: Pleased | 18
  Final: Could not be better | 0
  Final: Missing | 76

30. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: Do You Have Anyone You Would Call a Close Friend?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Yes | 113
  Baseline: No | 64
  Baseline: Missing | 67
  Final: Yes | 114
  Final: No | 58
  Final: Missing | 72

31. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: In the Last Week Have You Seen a Friend?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Yes | 87
  Baseline: No | 86
  Baseline: Missing | 71
  Final: Yes | 98
  Final: No | 72
  Final: Missing | 74

32. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With the Number and Quality of Your Friendships?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 3
  Baseline: Displeased | 45
  Baseline: Mostly dissatisfied | 37
  Baseline: Mixed | 31
  Baseline: Mostly satisfied | 36
  Baseline: Pleased | 23
  Baseline: Could not be better | 2
  Baseline: Missing | 67
  Final: Could not be worse | 3
  Final: Displeased | 23
  Final: Mostly dissatisfied | 35
  Final: Mixed | 36
  Final: Mostly satisfied | 50
  Final: Pleased | 26
  Final: Could not be better | 1
  Final: Missing | 70

33. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Leisure Activities?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 2
  Baseline: Displeased | 52
  Baseline: Mostly dissatisfied | 46
  Baseline: Mixed | 31
  Baseline: Mostly satisfied | 29
  Baseline: Pleased | 15
  Baseline: Could not be better | 2
  Baseline: Missing | 67
  Final: Could not be worse | 1
  Final: Displeased | 15
  Final: Mostly dissatisfied | 38
  Final: Mixed | 34
  Final: Mostly satisfied | 72
  Final: Pleased | 14
  Final: Could not be better | 0
  Final: Missing | 70

34. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Accomodation?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 4
  Baseline: Displeased | 31
  Baseline: Mostly dissatisfied | 24
  Baseline: Mixed | 26
  Baseline: Mostly satisfied | 41
  Baseline: Pleased | 46
  Baseline: Could not be better | 3
  Baseline: Missing | 69
  Final: Could not be worse | 1
  Final: Displeased | 15
  Final: Mostly dissatisfied | 17
  Final: Mixed | 38
  Final: Mostly satisfied | 45
  Final: Pleased | 51
  Final: Could not be better | 2
  Final: Missing | 75

35. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: In the Past Year, Have You Been Accused of a Crime?
Description: as for outcome 13
Time Frame: Baseline and final visit
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Yes | 4
  Baseline: No | 173
  Baseline: Missing | 67
  Final: Yes | 5
  Final: No | 170
  Final: Missing | 69

36. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: In the Past Year, Have You Been a Victim of Physical Violence?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Yes | 11
  Baseline: No | 165
  Baseline: Missing | 68
  Final: Yes | 9
  Final: No | 166
  Final: Missing | 69

37. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Personal Safety?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 6
  Baseline: Displeased | 34
  Baseline: Mostly dissatisfied | 27
  Baseline: Mixed | 45
  Baseline: Mostly satisfied | 30
  Baseline: Pleased | 27
  Baseline: Could not be better | 8
  Baseline: Missing | 67
  Final: Could not be worse | 2
  Final: Displeased | 11
  Final: Mostly dissatisfied | 14
  Final: Mixed | 33
  Final: Mostly satisfied | 63
  Final: Pleased | 45
  Final: Could not be better | 7
  Final: Missing | 69

38. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With the People You Live With?
Description: as for outcome 13
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 9
  Baseline: Displeased | 26
  Baseline: Mostly dissatisfied | 27
  Baseline: Mixed | 35
  Baseline: Mostly satisfied | 43
  Baseline: Pleased | 32
  Baseline: Could not be better | 4
  Baseline: Missing | 68
  Final: Could not be worse | 4
  Final: Displeased | 11
  Final: Mostly dissatisfied | 18
  Final: Mixed | 34
  Final: Mostly satisfied | 61
  Final: Pleased | 42
  Final: Could not be better | 4
  Final: Missing | 70

39. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Sex Life?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: The schizophrenia full analysis set included all subjects with a diagnosis of schizophrenia and who had received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 19
  Baseline: Displeased | 59
  Baseline: Mostly dissatisfied | 38
  Baseline: Mixed | 26
  Baseline: Mostly satisfied | 20
  Baseline: Pleased | 13
  Baseline: Could not be better | 1
  Baseline: Missing | 68
  Final: Could not be worse | 9
  Final: Displeased | 47
  Final: Mostly dissatisfied | 44
  Final: Mixed | 38
  Final: Mostly satisfied | 20
  Final: Pleased | 16
  Final: Could not be better | 0
  Final: Missing | 70

40. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Relationship With Your Family?
Description: as for outcome 2
Time Frame: Baseline and final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 3
  Baseline: Displeased | 29
  Baseline: Mostly dissatisfied | 32
  Baseline: Mixed | 38
  Baseline: Mostly satisfied | 41
  Baseline: Pleased | 30
  Baseline: Could not be better | 3
  Baseline: Missing | 68
  Final: Could not be worse | 1
  Final: Displeased | 11
  Final: Mostly dissatisfied | 20
  Final: Mixed | 40
  Final: Mostly satisfied | 58
  Final: Pleased | 43
  Final: Could not be better | 2
  Final: Missing | 69

41. Primary Outcome: Manchester Short Assessment of Quality of Life (MANSA) Scores (Schizophrenia Population) in Answer to: How Satisfied Are You With Your Health?
Description: as for outcome 2
Time Frame: Baseline to final visit (week 12)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  Baseline: Could not be worse | 4
  Baseline: Displeased | 31
  Baseline: Mostly dissatisfied | 27
  Baseline: Mixed | 36
  Baseline: Mostly satisfied | 40
  Baseline: Pleased | 37
  Baseline: Could not be better | 1
  Baseline: Missing | 68
  Final: Could not be worse | 0
  Final: Displeased | 18
  Final: Mostly dissatisfied | 14
  Final: Mixed | 26
  Final: Mostly satisfied | 66
  Final: Pleased | 50
  Final: Could not be better | 1
  Final: Missing | 69

42. Primary Outcome: Clinical Global Impression of Severity (CGI-S) Scores (Schizophrenia Population)
Description: as for outcome 1
Time Frame: Baseline
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 244
Participants
  (1) Normal, not ill | 1
  (2) Borderline mentally ill | 5
  (3) Mildly ill | 14
  (4) Moderately ill | 63
  (5) Absolutely clearly ill | 105
  (6) Severely ill | 33
  (7) Among the most severely ill subjects | 0
  Missing | 23

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 0/471
Other Adverse Events (participants affected / at risk) | 15/471
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=471)
Asthenia (General disorders) | 1
Condition aggrevated (General disorders) | 1
Fatigue (General disorders) | 3
Ill-defined disorder (General disorders) | 1
Rhinitis (Infections and infestations) | 1
Akathisia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 2
Extrapyramidal disorder (Nervous system disorders) | 4
Headache (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.